CLINICAL TRIAL: NCT01637805
Title: Phase 1 Study of Antigen-specific Cytotoxic T Lymphocytes Induced by Dendritic Cells Infected by Recombinant Adeno-associated Virus With CEA Gene in Stage IV Gastric Cancer
Brief Title: Clinical Safety and Preliminary Efficacy of AAV-DC-CTL Treatment in Stage IV Gastric Cancer
Acronym: AAV-DC-CTL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CIH-ZRP-201205001
Record Dates: First submitted 2012-07-03; First posted 2012-07-11 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2012-07

CONDITIONS: Stage IV Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

ARMS (1):
- AAV-DC-CTL (Experimental)
  Interventions: Biological: Antigen-specific cytotoxic T lymphocytes induced by dendritic cells infected by recombinant adeno-associated virus with CEA gene

INTERVENTIONS:
Biological: Antigen-specific cytotoxic T lymphocytes induced by dendritic cells infected by recombinant adeno-associated virus with CEA gene — AAV-DC-CTL: Intravenous infusion, 1×109 cells, day 14; one cycle every month; at least one cycle

SUMMARY:
The purpose of this study is to evaluate the clinical safety and preliminary efficacy of antigen-specific cytotoxic T lymphocytes induced by dendritic cells infected by recombinant adeno-associated virus with CEA gene in the treatment of stage IV gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Sex: male or female
* Age: from 18 to 80 years
* Histology: gastric cancer
* Clinical stage: stage IV
* Karnofsky performance status: more than 50%
* Expected survival: more than 2 months
* Sex: male or female
* Laboratory tests results 7 days before the start of treatment:

  * White blood cells: more than 3.0 × 109/L
  * Platelets: more than 100 × 109/L
  * Neutrophils: more than 1.5 × 109/L
  * Hemoglobin: more than 80g/L
  * Serum glutamate pyruvate transaminase: less than 2.5 folds of the upper normal limit (ULN)
  * Serum glutamic-oxal (o) acetic transaminase: less than 2.5 × ULN
  * Serum bilirubin: less than 1.25 × ULN
  * Serum creatinine: less than 1.25 × ULN
* Pregnancy test: the test of women of child-bearing period must be negative 7 days before the start of treatment
* Contraception: male and female subjects of child-bearing period must adopt a reliable method of contraception before entry into this study until 30 days after stopping this study
* Informed consent: subject must have the ability to understand and voluntarily sign a written informed consent

Exclusion Criteria:

* History of neoplasms: other neoplasms
* Medical history: mental disease, or congestive heart failure, or severe coronary artery disease, or cardiac arrhythmias, or concomitant corticosteroid therapy
* Metastasis: clinical symptoms of brain metastasis
* Other clinical trial: the subject received other clinical trial before this study
* Laboratory tests: the serum test of human immunodeficiency virus, or hepatitis B virus, or hepatitis C virus was positive
* Woman: pregnant or lactating women
* Compliance: poor compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-05; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 12 months
  CR + PR = ORR

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China